CLINICAL TRIAL: NCT02416596
Title: Routine Hysteroscopy in IVF/ICSI Cycles in Patients With Primary Unexplained Infertility: A Randomized Control Trial
Brief Title: Routine Hysteroscopy in IVF/ICSI Cycles in Patients With Primary Unexplained Infertility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Amr Abdulreheem, Dr, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ASMH-RH1
Record Dates: First submitted 2015-04-07; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Primary Infertility Unspecified; Infertility; Ovarian Hyperstimulation; Pregnancy
Keywords: ICSI; IVF; hysteroscopy; Supervision; In-vitro Fertilization
MeSH Terms: conditions — Infertility | interventions — Hysteroscopy; Hysteroscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Undergoing Hysterosopy (Experimental): This group will include 340 women with unexplained primary infertility undergoing their first trial of IVF/ICSI (intracytoplasmic sperm injection). This group will undergo hysteroscopy in the mid luteal phase of the proceeding cycle.
  Interventions: Procedure: Hysteroscopy; Device: Hysteroscope
- Group With No intervention (No Intervention): This group will include 340 women with unexplained primary infertility they will undergo their first trial of IVF/ICSI (intracytoplasmic sperm injection) without hysteroscopy in the mid Luteal phase of the proceeding cycle.

INTERVENTIONS:
Procedure: Hysteroscopy — Office hysteroscopy will be performed during the Luteal phase of the proceeding menstrual cycle.
  All OH (office hysteroscopy) procedures will be performed with a vaginoscopic approach without utilizing a speculum and applying traction to the cervix with a tenaculum.
  Antibiotic prophylaxis: None OH will be cancelled until after treatment of vaginal infection.
  Other Names: ROH: Routine Office Hysteroscopy
  Arms: Group Undergoing Hysterosopy
Device: Hysteroscope — The device used is a rigid hysteroscope (continuous flow, 30 degree forward oblique view) assembled in a 4-mm diameter diagnostic sheath with an atraumatic tip (Karl Storz Endoscopy).
  Illumination: High intensity cold light source and fiberoptic cable Distention medium: solution of 0.9% normal saline with pressure at 100-120 mmHg
  Arms: Group Undergoing Hysterosopy

SUMMARY:
The aim of the present study is to evaluate the impact of hysteroscopy prior to starting the IVF (in vitro fertilisation) cycle on treatment outcome in women with unexplained primary infertility.

DETAILED DESCRIPTION:
Proper history, examination and investigations are carried out to diagnose causes of infertility. Office hysteroscopy will be performed during the Luteal phase of the proceeding menstrual cycle using a rigid hysteroscope. Controlled ovarian hyper stimulation-embryo transfer (COH-ET) using the standard long protocol of induction used in Ain Shams University Maternity Hospitals ART (assisted reproductive techniques) unit.

Biochemical pregnancy will be determined by a positive pregnancy test performed 2 weeks after embryo transfer and clinical pregnancy will be defined by the presence of a gestational sac using transvaginal ultrasound performed 6 weeks after embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IVF/ICSI using the standard long GnRH-a (gonadotropin-releasing hormone-a) protocol.
* No evidence of uterine pathology by transvaginal ultrasound and hysterosalpingography during the follicular phase.
* Patients with unexplained primary infertility.

Exclusion Criteria:

* Patients undergoing IVF using other protocols of induction.
* Patients with evidence of uterine pathology by transvaginal ultrasound or hysterosalpingography during the follicular phase.
* Other causes of infertility rather than unexplained factor.
* Unexplained poor responders during the pending ICSI cycle.
* Patients with abnormal findings at hysteroscopy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 680 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Biochemical Pregnancy | 2-6 weeks
  Pregnancy determined by chemical test (2 weeks) and vag. U/S (ultrasound) (6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Khaled H Swaydan, PhD, Study Director — Ain Shams University (Obs&Gyn); Ahmed K Mekled, PhD, Study Chair — Ain Shams University (Obs&Gyn)

REFERENCES:
- [Background] El-Toukhy T, Sunkara SK, Coomarasamy A, Grace J, Khalaf Y. Outpatient hysteroscopy and subsequent IVF cycle outcome: a systematic review and meta-analysis. Reprod Biomed Online. 2008 May;16(5):712-9. doi: 10.1016/s1472-6483(10)60486-5. PMID 18492377
- [Background] Pundir J, Pundir V, Omanwa K, Khalaf Y, El-Toukhy T. Hysteroscopy prior to the first IVF cycle: a systematic review and meta-analysis. Reprod Biomed Online. 2014 Feb;28(2):151-61. doi: 10.1016/j.rbmo.2013.09.025. Epub 2013 Oct 5. PMID 24365027
- [Background] Loverro G, Nappi L, Vicino M, Carriero C, Vimercati A, Selvaggi L. Uterine cavity assessment in infertile women: comparison of transvaginal sonography and hysteroscopy. Eur J Obstet Gynecol Reprod Biol. 2001 Dec 10;100(1):67-71. doi: 10.1016/s0301-2115(01)00434-1. PMID 11728660
- [Background] Karayalcin R, Ozyer S, Ozcan S, Uzunlar O, Gurlek B, Moraloglu O, Batioglu S. Office hysteroscopy improves pregnancy rates following IVF. Reprod Biomed Online. 2012 Sep;25(3):261-6. doi: 10.1016/j.rbmo.2012.05.013. Epub 2012 Jun 16. PMID 22818094
- [Background] De Placido G, Clarizia R, Cadente C, Castaldo G, Romano C, Mollo A, Alviggi C, Conforti S. Compliance and diagnostic efficacy of mini-hysteroscopy versus traditional hysteroscopy in infertility investigation. Eur J Obstet Gynecol Reprod Biol. 2007 Nov;135(1):83-7. doi: 10.1016/j.ejogrb.2007.02.028. Epub 2007 May 3. PMID 17481803
- [Background] Almog B, Shalom-Paz E, Dufort D, Tulandi T. Promoting implantation by local injury to the endometrium. Fertil Steril. 2010 Nov;94(6):2026-9. doi: 10.1016/j.fertnstert.2009.12.075. Epub 2010 Feb 19. PMID 20171615
- [Background] Barash A, Dekel N, Fieldust S, Segal I, Schechtman E, Granot I. Local injury to the endometrium doubles the incidence of successful pregnancies in patients undergoing in vitro fertilization. Fertil Steril. 2003 Jun;79(6):1317-22. doi: 10.1016/s0015-0282(03)00345-5. PMID 12798877
- [Background] Bosteels J, Weyers S, Puttemans P, Panayotidis C, Van Herendael B, Gomel V, Mol BW, Mathieu C, D'Hooghe T. The effectiveness of hysteroscopy in improving pregnancy rates in subfertile women without other gynaecological symptoms: a systematic review. Hum Reprod Update. 2010 Jan-Feb;16(1):1-11. doi: 10.1093/humupd/dmp033. PMID 19744944
- [Background] Huang LN, Tan J, Hitkari J, Dahan MH. Should IVF be used as first-line treatment or as a last resort? A debate presented at the 2013 Canadian Fertility and Andrology Society meeting. Reprod Biomed Online. 2015 Feb;30(2):128-36. doi: 10.1016/j.rbmo.2014.10.004. Epub 2014 Oct 14. PMID 25498596
- [Background] Hughes E, Brown J, Collins JJ, Vanderkerchove P. Clomiphene citrate for unexplained subfertility in women. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD000057. doi: 10.1002/14651858.CD000057.pub2. PMID 20091498
- [Background] Lea RG, Sandra O. Immunoendocrine aspects of endometrial function and implantation. Reproduction. 2007 Sep;134(3):389-404. doi: 10.1530/REP-07-0167. PMID 17709558